CLINICAL TRIAL: NCT06545877
Title: REKOVELLE® PEN S.C. Injection 12μg/36μg/72μg for Controlled Ovarian Stimulation in Assisted Reproductive Technologies - General Drug Use-results Survey
Brief Title: REKOVELLE PEN for S.C. Injection General Drug Use Survey (Controlled Ovarian Stimulation in Assisted Reproductive Technologies)
Status: Recruiting | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000409
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This survey targets controlled ovarian stimulation with this drug for the development of multiple oocytes in women undergoing assisted reproduction (ART) such as in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI).

ELIGIBILITY:
Inclusion Criteria:

* Participants who received the REKOVELLE in controlled ovarian stimulation in assisted reproductive technologies and have consented to participate in the survey.

Exclusion Criteria:

* No exclusion criteria because data are collected under conditions of use in daily practice.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Women who are undergoing assisted reproduction (ART) such as in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2029-06-22 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | From initiation of the administration, in case of embryo transfer is not performed, until 1 week after oocyte collection, and in case embryo transfer is performed, 6 weeks after embryo transfer
  Frequency of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Ferring Investigational Site, Omitama, Ibaraki, Japan

IPD SHARING:
Plan to Share IPD: No